CLINICAL TRIAL: NCT00327860
Title: Chronic Kidney Disease in Children Prospective Cohort Study (CKiD)
Acronym: CKiD
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK66116; U01DK066143 (NIH); U01DK066174 (NIH); U24DK066116 (NIH); U24DK137522 (NIH); IRB10007880 (Other: CHOP IRB); IRB00011050 (Other: JHSPH IRB)
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine specimens were collected at the baseline visit and will be collected at each annual follow-up visit. Nail clippings and hair samples were collected at baseline. Whole blood samples were collected at baseline and processed to create immortalized cell lines, and DNA samples. Genetic and biological specimens will be stored at the NIDDK Central Repository, which is Precision for Medicine in Frederick, MD.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Cohort 1: Age between 1 and 16 years (before 17th birthday) and estimated (based on SCr) Schwartz GFR between 30 and 90 ml/min|1.73m2
- Cohort 2: Age between 1 and 16 years (before 17th birthday), estimated GFR between 45 and 90 ml/min|1.73m2 based on the updated Schwartz formula, and an equal distribution of children with glomerular and non-glomerular causes of disease were enrolled (i.e., 150 within each) and the study placed an upper limit of 60% for the percent of enrolled with non-glomerular disease.
- Cohort 3: Age between 6 months and 16 years (before 17th birthday) with non-glomerular diagnosis and duration of kidney disease less than 5 years will be enrolled.
- Cohort 4: Age between 16 and 22 years (before 23rd birthday) with moderately impaired kidney function as defined by estimated GFR less than 60 ml/min|1.73m2 based on U25eGFR OR individuals who have initiated kidney replacement therapy (dialysis or transplant).

SUMMARY:
The Division of Kidney, Urologic, and Hematologic Diseases (DKUHD) of the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), in collaboration with the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) and the National Heart, Lung and Blood Institute (NHLBI) funded a cooperative agreement including two Clinical Coordinating Centers (at Children's Hospital of Philadelphia and at Children's Mercy Hospital in Kansas City), a central biochemistry laboratory (at the University of Minnesota) and a Data Coordinating Center (at Johns Hopkins School of Public Health) to conduct a prospective epidemiological study of children with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
Since its inception in 2003, the scientific aims of CKiD have been to determine the risk factors for decline in kidney function and to define how progressive decline in kidney function impacts biomarkers of risk factors for cardiovascular disease; neurocognitive function and behavior; and growth failure and its associated morbidity.

The goals have been extended to understand the impact of childhood CKD on: the risk factors for decline in kidney function in childhood and young adulthood; the development of cardiovascular disease in adolescence and young adulthood; the trajectories of markers of metabolic bone disease and the relationship to cardiovascular endpoints; and the social function, neurocognitive function and emotional well-being of adolescents and young adults and the relationship to successful transfer to adult nephrology care.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 16 years (before 17th birthday) for Cohorts 1 and 2; age between 6 months and 16 years (before 17th birthday) for Cohort 3; age between 16 to 22 years (before 23rd birthday) for Cohort 4 and regularly seen by pediatric nephrologist prior to enrollment
* Estimated (based on SCr) Schwartz GFR between 30 and 90 ml/min|1.73m2 for Cohort 1 OR an estimated GFR between 45 and 90 ml/min|1.73m2 based on the updated Schwartz formula for Cohort 2; an estimated GFR ≤60 based on the CKiD Under 25 estimating equation (U25eGFR) OR KRT experience (dialysis or transplant) for Cohort 4
* Willingness and ability to provide informed consent and assent
* For Cohort 3, children with non-glomerular diagnosis and duration of kidney disease less than 5 years will be enrolled.

Exclusion Criteria:

* Solid organ (other than kidney), bone marrow or stem cell transplantation
* Cancer diagnosis and receiving treatment or within 12 months post completion of treatment
* HIV diagnosis and receiving treatment or within 12 months post completion of treatment
* Current pregnancy or pregnancy within past twelve months
* Inability to complete major data collection procedures
* Not fluent in English or Spanish
* Plans to move out of area of any participating CKiD site (families can be transferred to another CKiD site if the family moves)
* Existing moderate to severe congenital structural heart disease
* Genetic syndromes involving the central nervous system (e.g., Downs syndrome)
* History of severe to profound intellectual disability (i.e., Intelligence Quotient (IQ)<40, significant impairment in adaptive function and/or inability to independently execute self-care skills)
* For cohort 3, children who are expected to receive renal replacement therapy within 6 months of date of enrollment will not be recruited

Ages: 6 Months to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The CKiD Study is a multi-center, prospective cohort study of children, adolescents and young adults with a history of mild to moderate impaired kidney function. The study population consist of four cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2003-10 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Time to Kidney Replacement Therapy | Annually up to 5 years
  The time to Kidney Replacement Therapy (KRT) is assessed as the date of diagnosis to the date of KRT. The exact KRT date is self-reported by the participant and confirmed by medical record abstraction.

SECONDARY OUTCOMES:
Decline in Glomerular filtration rate (GFR) ml/min | Up to 25 years
  Define and identify novel and traditional risk factors for the accelerated decline of GFR at regular annual study visits.
Decline in GFR and risk of cardiovascular disease progression | Up to 25 years
  Analyze the association between decline in GFR and risk of progression of cardiovascular disease at regular annual study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Furth, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia; Bradley Warady, MD, Principal Investigator — Children's Mercy Kansas City; George Schwartz, MD, Principal Investigator — University of Rochester; Derek Ng, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Jesse Seegmiller, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Children's Mercy Kansas City, Kansas City, Missouri
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Thomas E, Klomhaus AM, Laster ML, Furth SL, Warady BA, Salusky IB, Hanudel MR. Associations between anemia and FGF23 in the CKiD study. Pediatr Nephrol. 2024 Mar;39(3):837-847. doi: 10.1007/s00467-023-06160-0. Epub 2023 Sep 26. PMID 37752381
- [Background] Sandokji I, Xu Y, Denburg M, Furth S, Abraham AG, Greenberg JH. Current and Novel Biomarkers of Progression Risk in Children with Chronic Kidney Disease. Nephron. 2024;148(1):1-10. doi: 10.1159/000530918. Epub 2023 May 15. PMID 37232009
- [Background] Ren X, Chen J, Abraham AG, Xu Y, Siewe A, Warady BA, Kimmel PL, Vasan RS, Rhee EP, Furth SL, Coresh J, Denburg M, Rebholz CM; Chronic Kidney Disease Biomarkers Consortium. Plasma Metabolomics of Dietary Intake of Protein-Rich Foods and Kidney Disease Progression in Children. J Ren Nutr. 2024 Mar;34(2):95-104. doi: 10.1053/j.jrn.2023.10.007. Epub 2023 Nov 8. PMID 37944769
- [Background] Lee AM, Xu Y, Hu J, Xiao R, Hooper SR, Hartung EA, Coresh J, Rhee EP, Vasan RS, Kimmel PL, Warady BA, Furth SL, Denburg MR; CKD Biomarkers Consortium. Longitudinal Plasma Metabolome Patterns and Relation to Kidney Function and Proteinuria in Pediatric CKD. Clin J Am Soc Nephrol. 2024 Jul 1;19(7):837-850. doi: 10.2215/CJN.0000000000000463. Epub 2024 May 6. PMID 38709558
- [Background] Lee AM, Xu Y, Hooper SR, Abraham AG, Hu J, Xiao R, Matheson MB, Brunson C, Rhee EP, Coresh J, Vasan RS, Schrauben S, Kimmel PL, Warady BA, Furth SL, Hartung EA, Denburg MR; CKD Biomarkers Consortium. Circulating Metabolomic Associations with Neurocognitive Outcomes in Pediatric CKD. Clin J Am Soc Nephrol. 2024 Jan 1;19(1):13-25. doi: 10.2215/CJN.0000000000000318. Epub 2023 Oct 23. PMID 37871960
- [Background] Inker LA, Tighiouart H, Adingwupu OM, Ng DK, Estrella MM, Maahs D, Yang W, Froissart M, Mauer M, Kalil R, Torres V, de Borst M, Klintmalm G, Poggio ED, Seegmiller JC, Rossing P, Furth SL, Warady BA, Schwartz GJ, Velez R, Coresh J, Levey AS. Performance of GFR Estimating Equations in Young Adults. Am J Kidney Dis. 2024 Feb;83(2):272-276. doi: 10.1053/j.ajkd.2023.06.008. Epub 2023 Sep 17. No abstract available. PMID 37717845
- [Background] Jiang K, Greenberg JH, Abraham A, Xu Y, Schelling JR, Feldman HI, Schrauben SJ, Waikar SS, Shlipak MG, Wettersten N, Coca SG, Vasan RS, Gutierrez OM, Ix JH, Warady BA, Kimmel PL, Bonventre JV, Parikh CR, Mitsnefes MM, Denburg MR, Furth S; CKD Biomarkers Consortium. Associations of Biomarkers of Kidney Tubule Health, Injury, and Inflammation with Left Ventricular Hypertrophy in Children with CKD. Kidney360. 2023 Aug 1;4(8):1039-1047. doi: 10.34067/KID.0000000000000183. Epub 2023 Jun 12. PMID 37303083
- [Background] Furth SL, Cole SR, Moxey-Mims M, Kaskel F, Mak R, Schwartz G, Wong C, Munoz A, Warady BA. Design and methods of the Chronic Kidney Disease in Children (CKiD) prospective cohort study. Clin J Am Soc Nephrol. 2006 Sep;1(5):1006-15. doi: 10.2215/CJN.01941205. Epub 2006 Jul 19. PMID 17699320
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- [Background] Schwartz GJ, Kwong T, Erway B, Warady B, Sokoll L, Hellerstein S, Dharnidharka V, Furth S, Munoz A. Validation of creatinine assays utilizing HPLC and IDMS traceable standards in sera of children. Pediatr Nephrol. 2009 Jan;24(1):113-9. doi: 10.1007/s00467-008-0957-0. Epub 2008 Sep 4. PMID 18769945
- [Background] Abraham AG, Schwartz GJ, Furth S, Warady BA, Munoz A. Longitudinal formulas to estimate GFR in children with CKD. Clin J Am Soc Nephrol. 2009 Nov;4(11):1724-30. doi: 10.2215/CJN.01860309. Epub 2009 Sep 17. PMID 19808217
- [Background] Schwartz GJ, Abraham AG, Furth SL, Warady BA, Munoz A. Optimizing iohexol plasma disappearance curves to measure the glomerular filtration rate in children with chronic kidney disease. Kidney Int. 2010 Jan;77(1):65-71. doi: 10.1038/ki.2009.398. PMID 19847157
- [Background] Checkley W, Brower RG, Munoz A; NIH Acute Respiratory Distress Syndrome Network Investigators. Inference for mutually exclusive competing events through a mixture of generalized gamma distributions. Epidemiology. 2010 Jul;21(4):557-65. doi: 10.1097/EDE.0b013e3181e090ed. PMID 20502337
- [Background] Abraham AG, Munoz A, Furth SL, Warady B, Schwartz GJ. Extracellular volume and glomerular filtration rate in children with chronic kidney disease. Clin J Am Soc Nephrol. 2011 Apr;6(4):741-7. doi: 10.2215/CJN.08020910. Epub 2011 Mar 24. PMID 21441126
- [Background] Copelovitch L, Warady BA, Furth SL. Insights from the Chronic Kidney Disease in Children (CKiD) study. Clin J Am Soc Nephrol. 2011 Aug;6(8):2047-53. doi: 10.2215/CJN.10751210. Epub 2011 Jul 22. PMID 21784815
- [Background] Fadrowski JJ, Neu AM, Schwartz GJ, Furth SL. Pediatric GFR estimating equations applied to adolescents in the general population. Clin J Am Soc Nephrol. 2011 Jun;6(6):1427-35. doi: 10.2215/CJN.06460710. Epub 2011 May 12. PMID 21566103
- [Background] Ng DK, Schwartz GJ, Jacobson LP, Palella FJ, Margolick JB, Warady BA, Furth SL, Munoz A. Universal GFR determination based on two time points during plasma iohexol disappearance. Kidney Int. 2011 Aug;80(4):423-30. doi: 10.1038/ki.2011.155. Epub 2011 Jun 8. PMID 21654718
- [Background] Pierce CB, Cox C, Saland JM, Furth SL, Munoz A. Methods for characterizing differences in longitudinal glomerular filtration rate changes between children with glomerular chronic kidney disease and those with nonglomerular chronic kidney disease. Am J Epidemiol. 2011 Sep 1;174(5):604-12. doi: 10.1093/aje/kwr121. Epub 2011 Aug 9. PMID 21828368
- [Background] Schwartz GJ, Schneider MF, Maier PS, Moxey-Mims M, Dharnidharka VR, Warady BA, Furth SL, Munoz A. Improved equations estimating GFR in children with chronic kidney disease using an immunonephelometric determination of cystatin C. Kidney Int. 2012 Aug;82(4):445-53. doi: 10.1038/ki.2012.169. PMID 22622496
- [Background] Wong CJ, Moxey-Mims M, Jerry-Fluker J, Warady BA, Furth SL. CKiD (CKD in children) prospective cohort study: a review of current findings. Am J Kidney Dis. 2012 Dec;60(6):1002-11. doi: 10.1053/j.ajkd.2012.07.018. Epub 2012 Sep 28. PMID 23022429
- [Background] Wuttke M, Schaefer F, Wong CS, Kottgen A. Genome-wide association studies in nephrology: using known associations for data checks. Am J Kidney Dis. 2015 Feb;65(2):217-22. doi: 10.1053/j.ajkd.2014.09.019. Epub 2014 Nov 18. PMID 25465167
- [Background] Wuttke M, Wong CS, Wuhl E, Epting D, Luo L, Hoppmann A, Doyon A, Li Y; CKDGen Consortium; Sozeri B, Thurn D, Helmstadter M, Huber TB, Blydt-Hansen TD, Kramer-Zucker A, Mehls O, Melk A, Querfeld U, Furth SL, Warady BA, Schaefer F, Kottgen A. Genetic loci associated with renal function measures and chronic kidney disease in children: the Pediatric Investigation for Genetic Factors Linked with Renal Progression Consortium. Nephrol Dial Transplant. 2016 Feb;31(2):262-9. doi: 10.1093/ndt/gfv342. Epub 2015 Sep 28. PMID 26420894
- [Background] Woroniecki RP, Ng DK, Limou S, Winkler CA, Reidy KJ, Mitsnefes M, Sampson MG, Wong CS, Warady BA, Furth SL, Kopp JB, Kaskel FJ. Renal and Cardiovascular Morbidities Associated with APOL1 Status among African-American and Non-African-American Children with Focal Segmental Glomerulosclerosis. Front Pediatr. 2016 Nov 17;4:122. doi: 10.3389/fped.2016.00122. eCollection 2016. PMID 27900314
- [Background] Ng DK, Schwartz GJ, Warady BA, Furth SL, Munoz A. Relationships of Measured Iohexol GFR and Estimated GFR With CKD-Related Biomarkers in Children and Adolescents. Am J Kidney Dis. 2017 Sep;70(3):397-405. doi: 10.1053/j.ajkd.2017.03.019. Epub 2017 May 24. PMID 28549535
- [Background] Schwartz GJ, Wang H, Erway B, Nordin G, Seegmiller J, Lieske JC, Back SE, Miller WG, Eckfeldt JH. Multicenter Laboratory Comparison of Iohexol Measurement. J Appl Lab Med. 2018 Mar;2(5):711-724. doi: 10.1373/jalm.2017.024240. PMID 31276084
- [Background] Wong CS, Kogon AJ, Warady BA, Furth SL, Lantos JD, Wilfond BS. Ethical and Policy Considerations for Genomic Testing in Pediatric Research: The Path Toward Disclosing Individual Research Results. Am J Kidney Dis. 2019 Jun;73(6):837-845. doi: 10.1053/j.ajkd.2019.01.020. Epub 2019 Mar 14. PMID 30879919
- [Background] Schwartz GJ, Cox C, Seegmiller JC, Maier PS, DiManno D, Furth SL, Warady BA, Munoz A. Recalibration of cystatin C using standardized material in Siemens nephelometers. Pediatr Nephrol. 2020 Feb;35(2):279-285. doi: 10.1007/s00467-019-04389-2. Epub 2019 Nov 3. PMID 31680199
- [Background] Furth S, Warady BA. Biomarkers, Imaging and Patient Reported Outcomes in The Chronic Kidney Disease in Children Study. Semin Nephrol. 2021 Sep;41(5):403-404. doi: 10.1016/j.semnephrol.2021.09.001. No abstract available. PMID 34916000
- [Background] Verbitsky M, Krishnamurthy S, Krithivasan P, Hughes D, Khan A, Marasa M, Vena N, Khosla P, Zhang J, Lim TY, Glessner JT, Weng C, Shang N, Shen Y, Hripcsak G, Hakonarson H, Ionita-Laza I, Levy B, Kenny EE, Loos RJF, Kiryluk K, Sanna-Cherchi S, Crosslin DR, Furth S, Warady BA, Igo RP Jr, Iyengar SK, Wong CS, Parsa A, Feldman HI, Gharavi AG. Genomic Disorders in CKD across the Lifespan. J Am Soc Nephrol. 2023 Apr 1;34(4):607-618. doi: 10.1681/ASN.2022060725. Epub 2022 Oct 27. PMID 36302597
- [Background] Fino NF, Adingwupu OM, Coresh J, Greene T, Haaland B, Shlipak MG, Costa E Silva VT, Kalil R, Mindikoglu AL, Furth SL, Seegmiller JC, Levey AS, Inker LA. Evaluation of novel candidate filtration markers from a global metabolomic discovery for glomerular filtration rate estimation. Kidney Int. 2024 Mar;105(3):582-592. doi: 10.1016/j.kint.2023.11.007. Epub 2023 Nov 23. PMID 38006943
- [Background] Menon G, Pierce CB, Ng DK; CKiD Study Investigators. Revisiting the Application of an Adult Kidney Failure Risk Prediction Equation to Children With CKD. Am J Kidney Dis. 2023 Jun;81(6):734-737. doi: 10.1053/j.ajkd.2022.11.004. Epub 2022 Dec 28. No abstract available. PMID 36586560
- [Background] Ng DK, Matheson MB, Schwartz GJ, Wang FM, Mendley SR, Furth SL, Warady BA; CKiD investigators. Development of an adaptive clinical web-based prediction tool for kidney replacement therapy in children with chronic kidney disease. Kidney Int. 2023 Nov;104(5):985-994. doi: 10.1016/j.kint.2023.06.020. Epub 2023 Jun 28. PMID 37391041
- [Background] Ng DK, Patel A, Cox C. Data quality control in longitudinal epidemiologic studies: conditional studentized residuals from linear mixed effects models for outlier detection in the setting of pediatric chronic kidney disease. Ann Epidemiol. 2023 Sep;85:38-44. doi: 10.1016/j.annepidem.2023.07.005. Epub 2023 Jul 16. PMID 37454831
- [Result] Ward RC, Kogon AJ, Matheson MB, Dawson A, Hooper SR, Molitor S, Wong C, Furth SL, Warady BA, Harshman LA. Psychotropic Medication Usage in Pediatric CKD: Reporting from the CKD in Children Cohort. Kidney360. 2024 Jul 1;5(7):967-973. doi: 10.34067/KID.0000000000000462. Epub 2024 May 13. PMID 38739451
- [Result] Ng DK, Munoz A; CKiD Study Investigators. Assessing bias in GFR estimating equations: improper GFR stratification can yield misleading results. Pediatr Nephrol. 2024 Jul;39(7):2139-2145. doi: 10.1007/s00467-024-06318-4. Epub 2024 Feb 24. PMID 38396091
- [Result] Kula AJ, Xu Y, Hill GD, Furth SL, Warady BA, Ng DK, Seegmiller J, Mitsnefes M; CKiD Study Investigators. Hypertension and Left Ventricular Strain in Pediatric Chronic Kidney Disease. Hypertension. 2024 Oct;81(10):2181-2188. doi: 10.1161/HYPERTENSIONAHA.124.23167. Epub 2024 Aug 28. PMID 39193718
- [Result] Kim HS, Ng DK, Matheson MB, Atkinson MA, Akhtar Y, Warady BA, Furth SL, Ruebner RL. Pubertal luteinizing hormone levels in children with chronic kidney disease and association with change in glomerular filtration rate. Pediatr Nephrol. 2024 May;39(5):1543-1549. doi: 10.1007/s00467-023-06210-7. Epub 2023 Nov 23. PMID 37996757
- [Result] Singh NS, Johnson RJ, Matheson MB, Carlson J, Hooper SR, Warady BA. A longitudinal analysis of the effect of anemia on executive functions in children with mild to moderate chronic kidney disease. Pediatr Nephrol. 2023 Mar;38(3):829-837. doi: 10.1007/s00467-022-05682-3. Epub 2022 Jul 21. PMID 35861871
- [Result] Kurzinski KL, Xu Y, Ng DK, Furth SL, Schwartz GJ, Warady BA; CKiD Study Investigators. Hyperkalemia in pediatric chronic kidney disease. Pediatr Nephrol. 2023 Sep;38(9):3083-3090. doi: 10.1007/s00467-023-05912-2. Epub 2023 Mar 20. PMID 36939915
- [Result] Brown DD, Roem J, Ng DK, Coghlan RF, Johnstone B, Horton W, Furth SL, Warady BA, Melamed ML, Dauber A; CKiD Study Investigators. Associations between collagen X biomarker and linear growth velocity in a pediatric chronic kidney disease cohort. Pediatr Nephrol. 2023 Dec;38(12):4145-4156. doi: 10.1007/s00467-023-06047-0. Epub 2023 Jul 19. PMID 37466864
- [Result] Schwartz GJ, Furth S, Cole SR, Warady B, Munoz A. Glomerular filtration rate via plasma iohexol disappearance: pilot study for chronic kidney disease in children. Kidney Int. 2006 Jun;69(11):2070-7. doi: 10.1038/sj.ki.5000385. PMID 16612328
- [Result] Flynn JT, Mitsnefes M, Pierce C, Cole SR, Parekh RS, Furth SL, Warady BA; Chronic Kidney Disease in Children Study Group. Blood pressure in children with chronic kidney disease: a report from the Chronic Kidney Disease in Children study. Hypertension. 2008 Oct;52(4):631-7. doi: 10.1161/HYPERTENSIONAHA.108.110635. Epub 2008 Aug 25. PMID 18725579
- [Result] Fadrowski JJ, Pierce CB, Cole SR, Moxey-Mims M, Warady BA, Furth SL. Hemoglobin decline in children with chronic kidney disease: baseline results from the chronic kidney disease in children prospective cohort study. Clin J Am Soc Nephrol. 2008 Mar;3(2):457-62. doi: 10.2215/CJN.03020707. Epub 2008 Jan 30. PMID 18235140
- [Result] Wong CS, Pierce CB, Cole SR, Warady BA, Mak RH, Benador NM, Kaskel F, Furth SL, Schwartz GJ; CKiD Investigators. Association of proteinuria with race, cause of chronic kidney disease, and glomerular filtration rate in the chronic kidney disease in children study. Clin J Am Soc Nephrol. 2009 Apr;4(4):812-9. doi: 10.2215/CJN.01780408. Epub 2009 Mar 18. PMID 19297612
- [Result] Dodson JL, Cohn SE, Cox C, Hmiel PS, Wood E, Mattoo TK, Warady BA, Furth SL. Urinary incontinence in the CKiD cohort and health related quality of life. J Urol. 2009 Oct;182(4 Suppl):2007-14. doi: 10.1016/j.juro.2009.06.012. Epub 2009 Aug 20. PMID 19695588
- [Result] Saland JM, Pierce CB, Mitsnefes MM, Flynn JT, Goebel J, Kupferman JC, Warady BA, Furth SL; CKiD Investigators. Dyslipidemia in children with chronic kidney disease. Kidney Int. 2010 Dec;78(11):1154-63. doi: 10.1038/ki.2010.311. Epub 2010 Aug 25. PMID 20736985
- [Result] Roumelioti ME, Wentz A, Schneider MF, Gerson AC, Hooper S, Benfield M, Warady BA, Furth SL, Unruh ML. Sleep and fatigue symptoms in children and adolescents with CKD: a cross-sectional analysis from the chronic kidney disease in children (CKiD) study. Am J Kidney Dis. 2010 Feb;55(2):269-80. doi: 10.1053/j.ajkd.2009.09.021. Epub 2010 Jan 19. PMID 20034719
- [Result] Mitsnefes M, Flynn J, Cohn S, Samuels J, Blydt-Hansen T, Saland J, Kimball T, Furth S, Warady B; CKiD Study Group. Masked hypertension associates with left ventricular hypertrophy in children with CKD. J Am Soc Nephrol. 2010 Jan;21(1):137-44. doi: 10.1681/ASN.2009060609. Epub 2009 Nov 16. PMID 19917781
- [Result] Gerson AC, Wentz A, Abraham AG, Mendley SR, Hooper SR, Butler RW, Gipson DS, Lande MB, Shinnar S, Moxey-Mims MM, Warady BA, Furth SL. Health-related quality of life of children with mild to moderate chronic kidney disease. Pediatrics. 2010 Feb;125(2):e349-57. doi: 10.1542/peds.2009-0085. Epub 2010 Jan 18. PMID 20083528
- [Result] Atkinson MA, Pierce CB, Zack RM, Barletta GM, Yadin O, Mentser M, Warady BA, Furth SL. Hemoglobin differences by race in children with CKD. Am J Kidney Dis. 2010 Jun;55(6):1009-17. doi: 10.1053/j.ajkd.2009.12.040. Epub 2010 Apr 24. PMID 20418001
- [Result] Furth SL, Abraham AG, Jerry-Fluker J, Schwartz GJ, Benfield M, Kaskel F, Wong C, Mak RH, Moxey-Mims M, Warady BA. Metabolic abnormalities, cardiovascular disease risk factors, and GFR decline in children with chronic kidney disease. Clin J Am Soc Nephrol. 2011 Sep;6(9):2132-40. doi: 10.2215/CJN.07100810. Epub 2011 Aug 12. PMID 21841064
- [Result] Greenbaum LA, Munoz A, Schneider MF, Kaskel FJ, Askenazi DJ, Jenkins R, Hotchkiss H, Moxey-Mims M, Furth SL, Warady BA. The association between abnormal birth history and growth in children with CKD. Clin J Am Soc Nephrol. 2011 Jan;6(1):14-21. doi: 10.2215/CJN.08481109. Epub 2010 Oct 28. PMID 21030583
- [Result] Hooper SR, Gerson AC, Butler RW, Gipson DS, Mendley SR, Lande MB, Shinnar S, Wentz A, Matheson M, Cox C, Furth SL, Warady BA. Neurocognitive functioning of children and adolescents with mild-to-moderate chronic kidney disease. Clin J Am Soc Nephrol. 2011 Aug;6(8):1824-30. doi: 10.2215/CJN.09751110. Epub 2011 Jul 7. PMID 21737850
- [Result] Lande MB, Gerson AC, Hooper SR, Cox C, Matheson M, Mendley SR, Gipson DS, Wong C, Warady BA, Furth SL, Flynn JT. Casual blood pressure and neurocognitive function in children with chronic kidney disease: a report of the children with chronic kidney disease cohort study. Clin J Am Soc Nephrol. 2011 Aug;6(8):1831-7. doi: 10.2215/CJN.00810111. Epub 2011 Jun 23. PMID 21700829
- [Result] Lo MM, Salisbury S, Scherer PE, Furth SL, Warady BA, Mitsnefes MM. Serum adiponectin complexes and cardiovascular risk in children with chronic kidney disease. Pediatr Nephrol. 2011 Nov;26(11):2009-17. doi: 10.1007/s00467-011-1906-x. Epub 2011 May 8. PMID 21553321
- [Result] Thomas R, Sanna-Cherchi S, Warady BA, Furth SL, Kaskel FJ, Gharavi AG. HNF1B and PAX2 mutations are a common cause of renal hypodysplasia in the CKiD cohort. Pediatr Nephrol. 2011 Jun;26(6):897-903. doi: 10.1007/s00467-011-1826-9. Epub 2011 Mar 5. PMID 21380624
- [Result] Wilson AC, Schneider MF, Cox C, Greenbaum LA, Saland J, White CT, Furth S, Warady BA, Mitsnefes MM. Prevalence and correlates of multiple cardiovascular risk factors in children with chronic kidney disease. Clin J Am Soc Nephrol. 2011 Dec;6(12):2759-65. doi: 10.2215/CJN.03010311. Epub 2011 Oct 6. PMID 21980183
- [Result] Atkinson MA, Pierce CB, Fadrowski JJ, Benador NM, White CT, Turman MA, Pan CG, Abraham AG, Warady BA, Furth SL. Association between common iron store markers and hemoglobin in children with chronic kidney disease. Pediatr Nephrol. 2012 Dec;27(12):2275-83. doi: 10.1007/s00467-012-2266-x. Epub 2012 Jul 27. PMID 22836305
- [Result] Brady TM, Schneider MF, Flynn JT, Cox C, Samuels J, Saland J, White CT, Furth S, Warady BA, Mitsnefes M. Carotid intima-media thickness in children with CKD: results from the CKiD study. Clin J Am Soc Nephrol. 2012 Dec;7(12):1930-7. doi: 10.2215/CJN.03130312. Epub 2012 Sep 13. PMID 22977209
- [Result] Flynn JT, Pierce CB, Miller ER 3rd, Charleston J, Samuels JA, Kupferman J, Furth SL, Warady BA; Chronic Kidney Disease in Children Study Group. Reliability of resting blood pressure measurement and classification using an oscillometric device in children with chronic kidney disease. J Pediatr. 2012 Mar;160(3):434-440.e1. doi: 10.1016/j.jpeds.2011.08.071. Epub 2011 Nov 1. PMID 22048052
- [Result] Nehus E, Furth S, Warady B, Mitsnefes M. Correlates of resistin in children with chronic kidney disease: the chronic kidney disease in children cohort. J Pediatr. 2012 Aug;161(2):276-80. doi: 10.1016/j.jpeds.2012.01.055. Epub 2012 Mar 14. PMID 22421264
- [Result] Samuels J, Ng D, Flynn JT, Mitsnefes M, Poffenbarger T, Warady BA, Furth S; Chronic Kidney Disease in Children Study Group. Ambulatory blood pressure patterns in children with chronic kidney disease. Hypertension. 2012 Jul;60(1):43-50. doi: 10.1161/HYPERTENSIONAHA.111.189266. Epub 2012 May 14. PMID 22585950
- [Result] Al-Uzri A, Matheson M, Gipson DS, Mendley SR, Hooper SR, Yadin O, Rozansky DJ, Moxey-Mims M, Furth SL, Warady BA, Gerson AC; Chronic Kidney Disease in Children Study Group. The impact of short stature on health-related quality of life in children with chronic kidney disease. J Pediatr. 2013 Sep;163(3):736-41.e1. doi: 10.1016/j.jpeds.2013.03.016. Epub 2013 Apr 26. PMID 23628375
- [Result] Fadrowski JJ, Abraham AG, Navas-Acien A, Guallar E, Weaver VM, Furth SL. Blood lead level and measured glomerular filtration rate in children with chronic kidney disease. Environ Health Perspect. 2013 Aug;121(8):965-70. doi: 10.1289/ehp.1205164. Epub 2013 May 21. PMID 23694739
- [Result] Hidalgo G, Ng DK, Moxey-Mims M, Minnick ML, Blydt-Hansen T, Warady BA, Furth SL. Association of income level with kidney disease severity and progression among children and adolescents with CKD: a report from the Chronic Kidney Disease in Children (CKiD) Study. Am J Kidney Dis. 2013 Dec;62(6):1087-94. doi: 10.1053/j.ajkd.2013.06.013. Epub 2013 Aug 7. PMID 23932090
- [Result] Kogon AJ, Pierce CB, Cox C, Brady TM, Mitsnefes MM, Warady BA, Furth SL, Flynn JT. Nephrotic-range proteinuria is strongly associated with poor blood pressure control in pediatric chronic kidney disease. Kidney Int. 2014 Apr;85(4):938-44. doi: 10.1038/ki.2013.352. Epub 2013 Sep 18. PMID 24048375
- [Result] Kupferman JC, Aronson Friedman L, Cox C, Flynn J, Furth S, Warady B, Mitsnefes M; CKiD Study Group. BP control and left ventricular hypertrophy regression in children with CKD. J Am Soc Nephrol. 2014 Jan;25(1):167-74. doi: 10.1681/ASN.2012121197. Epub 2013 Sep 26. PMID 24071004
- [Result] Omoloja A, Jerry-Fluker J, Ng DK, Abraham AG, Furth S, Warady BA, Mitsnefes M. Secondhand smoke exposure is associated with proteinuria in children with chronic kidney disease. Pediatr Nephrol. 2013 Aug;28(8):1243-51. doi: 10.1007/s00467-013-2456-1. Epub 2013 Apr 13. PMID 23584848
- [Result] Akchurin OM, Schneider MF, Mulqueen L, Brooks ER, Langman CB, Greenbaum LA, Furth SL, Moxey-Mims M, Warady BA, Kaskel FJ, Skversky AL. Medication adherence and growth in children with CKD. Clin J Am Soc Nephrol. 2014 Sep 5;9(9):1519-25. doi: 10.2215/CJN.01150114. Epub 2014 Jun 26. PMID 24970873
- [Result] Abraham AG, Mak RH, Mitsnefes M, White C, Moxey-Mims M, Warady B, Furth SL. Protein energy wasting in children with chronic kidney disease. Pediatr Nephrol. 2014 Jul;29(7):1231-8. doi: 10.1007/s00467-014-2768-9. Epub 2014 Feb 7. PMID 24504731
- [Result] Atkinson MA, Kim JY, Roy CN, Warady BA, White CT, Furth SL. Hepcidin and risk of anemia in CKD: a cross-sectional and longitudinal analysis in the CKiD cohort. Pediatr Nephrol. 2015 Apr;30(4):635-43. doi: 10.1007/s00467-014-2991-4. Epub 2014 Nov 8. PMID 25380788
- [Result] Barletta GM, Flynn J, Mitsnefes M, Samuels J, Friedman LA, Ng D, Cox C, Poffenbarger T, Warady B, Furth S. Heart rate and blood pressure variability in children with chronic kidney disease: a report from the CKiD study. Pediatr Nephrol. 2014 Jun;29(6):1059-65. doi: 10.1007/s00467-013-2737-8. Epub 2014 Feb 2. PMID 24488505
- [Result] Blydt-Hansen TD, Pierce CB, Cai Y, Samsonov D, Massengill S, Moxey-Mims M, Warady BA, Furth SL. Medication treatment complexity and adherence in children with CKD. Clin J Am Soc Nephrol. 2014 Feb;9(2):247-54. doi: 10.2215/CJN.05750513. Epub 2013 Nov 21. PMID 24262500
- [Result] Flynn JT, Ng DK, Chan GJ, Samuels J, Furth S, Warady B, Greenbaum LA; Chronic Kidney Disease in Children Study. The effect of abnormal birth history on ambulatory blood pressure and disease progression in children with chronic kidney disease. J Pediatr. 2014 Jul;165(1):154-162.e1. doi: 10.1016/j.jpeds.2014.02.051. Epub 2014 Mar 31. PMID 24698454
- [Result] Hartung EA, Matheson M, Lande MB, Dell KM, Guay-Woodford LM, Gerson AC, Warady BA, Hooper SR, Furth SL. Neurocognition in children with autosomal recessive polycystic kidney disease in the CKiD cohort study. Pediatr Nephrol. 2014 Oct;29(10):1957-65. doi: 10.1007/s00467-014-2816-5. Epub 2014 May 15. PMID 24828609
- [Result] Mendley SR, Matheson MB, Shinnar S, Lande MB, Gerson AC, Butler RW, Warady BA, Furth SL, Hooper SR. Duration of chronic kidney disease reduces attention and executive function in pediatric patients. Kidney Int. 2015 Apr;87(4):800-6. doi: 10.1038/ki.2014.323. Epub 2014 Sep 24. PMID 25252026
- [Result] Mitsnefes M, Scherer PE, Friedman LA, Gordillo R, Furth S, Warady BA; CKiD study group. Ceramides and cardiac function in children with chronic kidney disease. Pediatr Nephrol. 2014 Mar;29(3):415-22. doi: 10.1007/s00467-013-2642-1. Epub 2014 Jan 5. PMID 24389650
- [Result] Portale AA, Wolf M, Juppner H, Messinger S, Kumar J, Wesseling-Perry K, Schwartz GJ, Furth SL, Warady BA, Salusky IB. Disordered FGF23 and mineral metabolism in children with CKD. Clin J Am Soc Nephrol. 2014 Feb;9(2):344-53. doi: 10.2215/CJN.05840513. Epub 2013 Dec 5. PMID 24311704
- [Result] Rodig NM, McDermott KC, Schneider MF, Hotchkiss HM, Yadin O, Seikaly MG, Furth SL, Warady BA. Growth in children with chronic kidney disease: a report from the Chronic Kidney Disease in Children Study. Pediatr Nephrol. 2014 Oct;29(10):1987-95. doi: 10.1007/s00467-014-2812-9. Epub 2014 Apr 12. PMID 24728472
- [Result] Zhong Y, Munoz A, Schwartz GJ, Warady BA, Furth SL, Abraham AG. Nonlinear trajectory of GFR in children before RRT. J Am Soc Nephrol. 2014 May;25(5):913-7. doi: 10.1681/ASN.2013050487. Epub 2014 Jan 2. PMID 24385591
- [Result] Fathallah-Shaykh SA, Flynn JT, Pierce CB, Abraham AG, Blydt-Hansen TD, Massengill SF, Moxey-Mims MM, Warady BA, Furth SL, Wong CS. Progression of pediatric CKD of nonglomerular origin in the CKiD cohort. Clin J Am Soc Nephrol. 2015 Apr 7;10(4):571-7. doi: 10.2215/CJN.07480714. Epub 2015 Jan 29. PMID 25635034
- [Result] Denburg MR, Kumar J, Jemielita T, Brooks ER, Skversky A, Portale AA, Salusky IB, Warady BA, Furth SL, Leonard MB. Fracture Burden and Risk Factors in Childhood CKD: Results from the CKiD Cohort Study. J Am Soc Nephrol. 2016 Feb;27(2):543-50. doi: 10.1681/ASN.2015020152. Epub 2015 Jul 2. PMID 26139439
- [Result] Kumar J, McDermott K, Abraham AG, Friedman LA, Johnson VL, Kaskel FJ, Furth SL, Warady BA, Portale AA, Melamed ML. Prevalence and correlates of 25-hydroxyvitamin D deficiency in the Chronic Kidney Disease in Children (CKiD) cohort. Pediatr Nephrol. 2016 Jan;31(1):121-9. doi: 10.1007/s00467-015-3190-7. Epub 2015 Aug 26. PMID 26307635
- [Result] Mitsnefes MM, Pierce C, Flynn J, Samuels J, Dionne J, Furth S, Warady B; CKiD study group. Can office blood pressure readings predict masked hypertension? Pediatr Nephrol. 2016 Jan;31(1):163-6. doi: 10.1007/s00467-015-3212-5. Epub 2015 Sep 28. PMID 26416480
- [Result] Rodenbach KE, Schneider MF, Furth SL, Moxey-Mims MM, Mitsnefes MM, Weaver DJ, Warady BA, Schwartz GJ. Hyperuricemia and Progression of CKD in Children and Adolescents: The Chronic Kidney Disease in Children (CKiD) Cohort Study. Am J Kidney Dis. 2015 Dec;66(6):984-92. doi: 10.1053/j.ajkd.2015.06.015. Epub 2015 Jul 21. PMID 26209544
- [Result] Verbitsky M, Sanna-Cherchi S, Fasel DA, Levy B, Kiryluk K, Wuttke M, Abraham AG, Kaskel F, Kottgen A, Warady BA, Furth SL, Wong CS, Gharavi AG. Genomic imbalances in pediatric patients with chronic kidney disease. J Clin Invest. 2015 May;125(5):2171-8. doi: 10.1172/JCI80877. Epub 2015 Apr 20. PMID 25893603
- [Result] Warady BA, Abraham AG, Schwartz GJ, Wong CS, Munoz A, Betoko A, Mitsnefes M, Kaskel F, Greenbaum LA, Mak RH, Flynn J, Moxey-Mims MM, Furth S. Predictors of Rapid Progression of Glomerular and Nonglomerular Kidney Disease in Children and Adolescents: The Chronic Kidney Disease in Children (CKiD) Cohort. Am J Kidney Dis. 2015 Jun;65(6):878-88. doi: 10.1053/j.ajkd.2015.01.008. Epub 2015 Mar 19. PMID 25799137
- [Result] Ayestaran FW, Schneider MF, Kaskel FJ, Srivaths PR, Seo-Mayer PW, Moxey-Mims M, Furth SL, Warady BA, Greenbaum LA. Perceived appetite and clinical outcomes in children with chronic kidney disease. Pediatr Nephrol. 2016 Jul;31(7):1121-7. doi: 10.1007/s00467-016-3321-9. Epub 2016 Feb 8. PMID 26857711
- [Result] Dell KM, Matheson M, Hartung EA, Warady BA, Furth SL; Chronic Kidney Disease in Children (CKiD) Study. Kidney Disease Progression in Autosomal Recessive Polycystic Kidney Disease. J Pediatr. 2016 Apr;171:196-201.e1. doi: 10.1016/j.jpeds.2015.12.079. Epub 2016 Jan 28. PMID 26831744
- [Result] Hooper SR, Gerson AC, Johnson RJ, Mendley SR, Shinnar S, Lande MB, Matheson MB, Gipson DS, Morgenstern B, Warady BA, Furth SL. Neurocognitive, Social-Behavioral, and Adaptive Functioning in Preschool Children with Mild to Moderate Kidney Disease. J Dev Behav Pediatr. 2016 Apr;37(3):231-8. doi: 10.1097/DBP.0000000000000267. PMID 26890559
- [Result] Kogon AJ, Matheson MB, Flynn JT, Gerson AC, Warady BA, Furth SL, Hooper SR; Chronic Kidney Disease in Children (CKiD) Study Group. Depressive Symptoms in Children with Chronic Kidney Disease. J Pediatr. 2016 Jan;168:164-170.e1. doi: 10.1016/j.jpeds.2015.09.040. Epub 2015 Oct 23. PMID 26505290
- [Result] Hartung EA, Dell KM, Matheson M, Warady BA, Furth SL. Growth in Children with Autosomal Recessive Polycystic Kidney Disease in the CKiD Cohort Study. Front Pediatr. 2016 Aug 10;4:82. doi: 10.3389/fped.2016.00082. eCollection 2016. PMID 27559537
- [Result] Lande MB, Mendley SR, Matheson MB, Shinnar S, Gerson AC, Samuels JA, Warady BA, Furth SL, Hooper SR. Association of blood pressure variability and neurocognition in children with chronic kidney disease. Pediatr Nephrol. 2016 Nov;31(11):2137-44. doi: 10.1007/s00467-016-3425-2. Epub 2016 Jun 5. PMID 27263021
- [Result] Ng DK, Moxey-Mims M, Warady BA, Furth SL, Munoz A. Racial differences in renal replacement therapy initiation among children with a nonglomerular cause of chronic kidney disease. Ann Epidemiol. 2016 Nov;26(11):780-787.e1. doi: 10.1016/j.annepidem.2016.09.011. Epub 2016 Oct 8. PMID 27789133
- [Result] Portale AA, Wolf MS, Messinger S, Perwad F, Juppner H, Warady BA, Furth SL, Salusky IB. Fibroblast Growth Factor 23 and Risk of CKD Progression in Children. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):1989-1998. doi: 10.2215/CJN.02110216. Epub 2016 Aug 25. PMID 27561289
- [Result] Ruebner RL, Ng D, Mitsnefes M, Foster BJ, Meyers K, Warady B, Furth SL. Cardiovascular Disease Risk Factors and Left Ventricular Hypertrophy in Girls and Boys With CKD. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):1962-1968. doi: 10.2215/CJN.01270216. Epub 2016 Sep 14. PMID 27630183
- [Result] Abraham AG, Betoko A, Fadrowski JJ, Pierce C, Furth SL, Warady BA, Munoz A. Renin-angiotensin II-aldosterone system blockers and time to renal replacement therapy in children with CKD. Pediatr Nephrol. 2017 Apr;32(4):643-649. doi: 10.1007/s00467-016-3512-4. Epub 2016 Nov 8. PMID 27826732
- [Result] Brady TM, Townsend K, Schneider MF, Cox C, Kimball T, Madueme P, Warady B, Furth S, Mitsnefes M. Cystatin C and Cardiac Measures in Children and Adolescents With CKD. Am J Kidney Dis. 2017 Feb;69(2):247-256. doi: 10.1053/j.ajkd.2016.08.036. Epub 2016 Nov 14. PMID 27856090
- [Result] Chen W, Ducharme-Smith K, Davis L, Hui WF, Warady BA, Furth SL, Abraham AG, Betoko A. Dietary sources of energy and nutrient intake among children and adolescents with chronic kidney disease. Pediatr Nephrol. 2017 Jul;32(7):1233-1241. doi: 10.1007/s00467-017-3580-0. Epub 2017 Feb 16. PMID 28210840
- [Result] Fuhrman DY, Schneider MF, Dell KM, Blydt-Hansen TD, Mak R, Saland JM, Furth SL, Warady BA, Moxey-Mims MM, Schwartz GJ. Albuminuria, Proteinuria, and Renal Disease Progression in Children with CKD. Clin J Am Soc Nephrol. 2017 Jun 7;12(6):912-920. doi: 10.2215/CJN.11971116. Epub 2017 May 25. PMID 28546440
- [Result] Hui WF, Betoko A, Savant JD, Abraham AG, Greenbaum LA, Warady B, Moxey-Mims MM, Furth SL. Assessment of dietary intake of children with chronic kidney disease. Pediatr Nephrol. 2017 Mar;32(3):485-494. doi: 10.1007/s00467-016-3491-5. Epub 2016 Sep 29. PMID 27687620
- [Result] Knight A, Kogon AJ, Matheson MB, Warady BA, Furth SL, Hooper SR. Cognitive Function in Children with Lupus Nephritis: A Cross-Sectional Comparison with Children with Other Glomerular Chronic Kidney Diseases. J Pediatr. 2017 Oct;189:181-188.e1. doi: 10.1016/j.jpeds.2017.06.044. Epub 2017 Jul 19. PMID 28734655
- [Result] Lopez-Rivera E, Liu YP, Verbitsky M, Anderson BR, Capone VP, Otto EA, Yan Z, Mitrotti A, Martino J, Steers NJ, Fasel DA, Vukojevic K, Deng R, Racedo SE, Liu Q, Werth M, Westland R, Vivante A, Makar GS, Bodria M, Sampson MG, Gillies CE, Vega-Warner V, Maiorana M, Petrey DS, Honig B, Lozanovski VJ, Salomon R, Heidet L, Carpentier W, Gaillard D, Carrea A, Gesualdo L, Cusi D, Izzi C, Scolari F, van Wijk JA, Arapovic A, Saraga-Babic M, Saraga M, Kunac N, Samii A, McDonald-McGinn DM, Crowley TB, Zackai EH, Drozdz D, Miklaszewska M, Tkaczyk M, Sikora P, Szczepanska M, Mizerska-Wasiak M, Krzemien G, Szmigielska A, Zaniew M, Darlow JM, Puri P, Barton D, Casolari E, Furth SL, Warady BA, Gucev Z, Hakonarson H, Flogelova H, Tasic V, Latos-Bielenska A, Materna-Kiryluk A, Allegri L, Wong CS, Drummond IA, D'Agati V, Imamoto A, Barasch JM, Hildebrandt F, Kiryluk K, Lifton RP, Morrow BE, Jeanpierre C, Papaioannou VE, Ghiggeri GM, Gharavi AG, Katsanis N, Sanna-Cherchi S. Genetic Drivers of Kidney Defects in the DiGeorge Syndrome. N Engl J Med. 2017 Feb 23;376(8):742-754. doi: 10.1056/NEJMoa1609009. Epub 2017 Jan 25. PMID 28121514
- [Result] Ng DK, Robertson CC, Woroniecki RP, Limou S, Gillies CE, Reidy KJ, Winkler CA, Hingorani S, Gibson KL, Hjorten R, Sethna CB, Kopp JB, Moxey-Mims M, Furth SL, Warady BA, Kretzler M, Sedor JR, Kaskel FJ, Sampson MG. APOL1-associated glomerular disease among African-American children: a collaboration of the Chronic Kidney Disease in Children (CKiD) and Nephrotic Syndrome Study Network (NEPTUNE) cohorts. Nephrol Dial Transplant. 2017 Jun 1;32(6):983-990. doi: 10.1093/ndt/gfw061. PMID 27190333
- [Result] Savant JD, Betoko A, Meyers KE, Mitsnefes M, Flynn JT, Townsend RR, Greenbaum LA, Dart A, Warady B, Furth SL. Vascular Stiffness in Children With Chronic Kidney Disease. Hypertension. 2017 May;69(5):863-869. doi: 10.1161/HYPERTENSIONAHA.116.07653. Epub 2017 Apr 3. PMID 28373588
- [Result] Verbitsky M, Kogon AJ, Matheson M, Hooper SR, Wong CS, Warady BA, Furth SL, Gharavi AG. Genomic Disorders and Neurocognitive Impairment in Pediatric CKD. J Am Soc Nephrol. 2017 Aug;28(8):2303-2309. doi: 10.1681/ASN.2016101108. Epub 2017 Mar 27. PMID 28348065
- [Result] Patel HP, Saland JM, Ng DK, Jiang S, Warady BA, Furth SL, Flynn JT. Waist Circumference and Body Mass Index in Children with Chronic Kidney Disease and Metabolic, Cardiovascular, and Renal Outcomes. J Pediatr. 2017 Dec;191:133-139. doi: 10.1016/j.jpeds.2017.08.047. PMID 29173296
- [Result] Barletta GM, Pierce C, Mitsnefes M, Samuels J, Warady BA, Furth S, Flynn J. Is Blood Pressure Improving in Children With Chronic Kidney Disease? A Period Analysis. Hypertension. 2018 Mar;71(3):444-450. doi: 10.1161/HYPERTENSIONAHA.117.09649. Epub 2018 Jan 2. PMID 29295853
- [Result] Brooks ER, Haymond S, Rademaker A, Pierce C, Helenowski I, Passman R, Vicente F, Warady BA, Furth SL, Langman CB. Contribution of symmetric dimethylarginine to GFR decline in pediatric chronic kidney disease. Pediatr Nephrol. 2018 Apr;33(4):697-704. doi: 10.1007/s00467-017-3842-x. Epub 2017 Dec 7. PMID 29214443
- [Result] Furth SL, Pierce C, Hui WF, White CA, Wong CS, Schaefer F, Wuhl E, Abraham AG, Warady BA; Chronic Kidney Disease in Children (CKiD); Effect of Strict Blood Pressure Control and ACE Inhibition on the Progression of CRF in Pediatric Patients (ESCAPE) Study Investigators. Estimating Time to ESRD in Children With CKD. Am J Kidney Dis. 2018 Jun;71(6):783-792. doi: 10.1053/j.ajkd.2017.12.011. Epub 2018 Apr 10. PMID 29653769
- [Result] Ku E, McCulloch CE, Warady BA, Furth SL, Grimes BA, Mitsnefes MM. Twenty-Four-Hour Ambulatory Blood Pressure versus Clinic Blood Pressure Measurements and Risk of Adverse Outcomes in Children with CKD. Clin J Am Soc Nephrol. 2018 Mar 7;13(3):422-428. doi: 10.2215/CJN.09630917. Epub 2018 Feb 13. PMID 29440119
- [Result] Lalan S, Jiang S, Ng DK, Kupferman F, Warady BA, Furth S, Mitsnefes MM. Cardiometabolic Risk Factors, Metabolic Syndrome, and Chronic Kidney Disease Progression in Children. J Pediatr. 2018 Nov;202:163-170. doi: 10.1016/j.jpeds.2018.06.007. Epub 2018 Jul 2. PMID 30041938
- [Result] Mitsnefes MM, Betoko A, Schneider MF, Salusky IB, Wolf MS, Juppner H, Warady BA, Furth SL, Portale AA. FGF23 and Left Ventricular Hypertrophy in Children with CKD. Clin J Am Soc Nephrol. 2018 Jan 6;13(1):45-52. doi: 10.2215/CJN.02110217. Epub 2017 Oct 12. PMID 29025789
- [Result] Ng DK, Portale AA, Furth SL, Warady BA, Munoz A. Time-varying coefficient of determination to quantify the explanatory power of biomarkers on longitudinal GFR among children with chronic kidney disease. Ann Epidemiol. 2018 Aug;28(8):549-556. doi: 10.1016/j.annepidem.2018.05.002. Epub 2018 May 17. PMID 29887227
- [Result] Ng DK, Schwartz GJ, Schneider MF, Furth SL, Warady BA. Combination of pediatric and adult formulas yield valid glomerular filtration rate estimates in young adults with a history of pediatric chronic kidney disease. Kidney Int. 2018 Jul;94(1):170-177. doi: 10.1016/j.kint.2018.01.034. Epub 2018 May 5. PMID 29735307
- [Result] Ricardo AC, Pereira LN, Betoko A, Goh V, Amarah A, Warady BA, Moxey-Mims M, Furth S, Lash JP; Chronic Kidney Disease in Children (CKiD) Cohort Investigators. Parental health literacy and progression of chronic kidney disease in children. Pediatr Nephrol. 2018 Oct;33(10):1759-1764. doi: 10.1007/s00467-018-3962-y. Epub 2018 Jun 14. PMID 29948310
- [Result] Sgambat K, Roem J, Mitsnefes M, Portale AA, Furth S, Warady B, Moudgil A. Waist-to-height ratio, body mass index, and cardiovascular risk profile in children with chronic kidney disease. Pediatr Nephrol. 2018 Sep;33(9):1577-1583. doi: 10.1007/s00467-018-3987-2. Epub 2018 Jun 5. PMID 29872963
- [Result] Altemose KE, Kumar J, Portale AA, Warady BA, Furth SL, Fadrowski JJ, Atkinson MA. Vitamin D insufficiency, hemoglobin, and anemia in children with chronic kidney disease. Pediatr Nephrol. 2018 Nov;33(11):2131-2136. doi: 10.1007/s00467-018-4020-5. Epub 2018 Jul 14. PMID 30008129
- [Result] Malits J, Attina TM, Karthikraj R, Kannan K, Naidu M, Furth S, Warady BA, Vento S, Trachtman H, Trasande L. Renal Function and exposure to Bisphenol A and phthalates in children with Chronic Kidney Disease. Environ Res. 2018 Nov;167:575-582. doi: 10.1016/j.envres.2018.08.006. Epub 2018 Aug 9. PMID 30172191
- [Result] Atkinson MA, Xiao R, Kottgen A, Wuhl E, Wong CS, Wuttke M, Bayazit AK, Caliskan S, Warady BA, Schaefer F, Furth SL. Genetic associations of hemoglobin in children with chronic kidney disease in the PediGFR Consortium. Pediatr Res. 2019 Feb;85(3):324-328. doi: 10.1038/s41390-018-0148-z. Epub 2018 Aug 15. PMID 30140068
- [Result] Brooks ER, Lin DC, Langman CB, Thompson JW, St John-Williams L, Furth SL, Warady B, Haymond S. Metabolomic Patterns in Adolescents With Mild to Moderate CKD. Kidney Int Rep. 2019 Jan 28;4(5):720-723. doi: 10.1016/j.ekir.2019.01.009. eCollection 2019 May. No abstract available. PMID 31080927
- [Result] Harshman LA, Johnson RJ, Matheson MB, Kogon AJ, Shinnar S, Gerson AC, Warady BA, Furth SL, Hooper SR. Academic achievement in children with chronic kidney disease: a report from the CKiD cohort. Pediatr Nephrol. 2019 Apr;34(4):689-696. doi: 10.1007/s00467-018-4144-7. Epub 2018 Nov 17. PMID 30448874
- [Result] Li Y, Greenbaum LA, Warady BA, Furth SL, Ng DK. Short stature in advanced pediatric CKD is associated with faster time to reduced kidney function after transplant. Pediatr Nephrol. 2019 May;34(5):897-905. doi: 10.1007/s00467-018-4165-2. Epub 2019 Jan 9. PMID 30627858
- [Result] Ng DK, Matheson MB, Warady BA, Mendley SR, Furth SL, Munoz A. Incidence of Initial Renal Replacement Therapy Over the Course of Kidney Disease in Children. Am J Epidemiol. 2019 Dec 31;188(12):2156-2164. doi: 10.1093/aje/kwz220. PMID 31595948
- [Result] Ruebner RL, Hooper SR, Parrish C, Furth SL, Fadrowski JJ. Environmental lead exposure is associated with neurocognitive dysfunction in children with chronic kidney disease. Pediatr Nephrol. 2019 Nov;34(11):2371-2379. doi: 10.1007/s00467-019-04306-7. Epub 2019 Jul 20. PMID 31327061
- [Result] Saland JM, Kupferman JC, Pierce CB, Flynn JT, Mitsnefes MM, Warady BA, Furth SL. Change in Dyslipidemia with Declining Glomerular Filtration Rate and Increasing Proteinuria in Children with CKD. Clin J Am Soc Nephrol. 2019 Dec 6;14(12):1711-1718. doi: 10.2215/CJN.03110319. Epub 2019 Nov 11. PMID 31712386
- [Result] Sethna CB, Ng DK, Jiang S, Saland J, Warady BA, Furth S, Meyers KE. Cardiovascular disease risk among children with focal segmental glomerulosclerosis: a report from the chronic kidney disease in children study. Pediatr Nephrol. 2019 Aug;34(8):1403-1412. doi: 10.1007/s00467-019-04229-3. Epub 2019 Mar 22. PMID 30903375
- [Result] Sgambat K, Matheson MB, Hooper SR, Warady B, Furth S, Moudgil A. Prevalence and outcomes of fragility: a frailty-inflammation phenotype in children with chronic kidney disease. Pediatr Nephrol. 2019 Dec;34(12):2563-2569. doi: 10.1007/s00467-019-04313-8. Epub 2019 Aug 2. PMID 31375914
- [Result] Staples A, Wong C, Schwartz GJ. Iohexol-measured glomerular filtration rate in children and adolescents with chronic kidney disease: a pilot study comparing venous and finger stick methods. Pediatr Nephrol. 2019 Mar;34(3):459-464. doi: 10.1007/s00467-018-4110-4. Epub 2018 Oct 12. PMID 30315406
- [Result] Verbitsky M, Westland R, Perez A, Kiryluk K, Liu Q, Krithivasan P, Mitrotti A, Fasel DA, Batourina E, Sampson MG, Bodria M, Werth M, Kao C, Martino J, Capone VP, Vivante A, Shril S, Kil BH, Marasa M, Zhang JY, Na YJ, Lim TY, Ahram D, Weng PL, Heinzen EL, Carrea A, Piaggio G, Gesualdo L, Manca V, Masnata G, Gigante M, Cusi D, Izzi C, Scolari F, van Wijk JAE, Saraga M, Santoro D, Conti G, Zamboli P, White H, Drozdz D, Zachwieja K, Miklaszewska M, Tkaczyk M, Tomczyk D, Krakowska A, Sikora P, Jarmolinski T, Borszewska-Kornacka MK, Pawluch R, Szczepanska M, Adamczyk P, Mizerska-Wasiak M, Krzemien G, Szmigielska A, Zaniew M, Dobson MG, Darlow JM, Puri P, Barton DE, Furth SL, Warady BA, Gucev Z, Lozanovski VJ, Tasic V, Pisani I, Allegri L, Rodas LM, Campistol JM, Jeanpierre C, Alam S, Casale P, Wong CS, Lin F, Miranda DM, Oliveira EA, Simoes-E-Silva AC, Barasch JM, Levy B, Wu N, Hildebrandt F, Ghiggeri GM, Latos-Bielenska A, Materna-Kiryluk A, Zhang F, Hakonarson H, Papaioannou VE, Mendelsohn CL, Gharavi AG, Sanna-Cherchi S. The copy number variation landscape of congenital anomalies of the kidney and urinary tract. Nat Genet. 2019 Jan;51(1):117-127. doi: 10.1038/s41588-018-0281-y. Epub 2018 Dec 21. PMID 30578417
- [Result] Atkinson MA, Roem JL, Gajjar A, Warady BA, Furth SL, Munoz A. Mode of initial renal replacement therapy and transplant outcomes in the chronic kidney disease in children (CKiD) study. Pediatr Nephrol. 2020 Jun;35(6):1015-1021. doi: 10.1007/s00467-019-04416-2. Epub 2019 Dec 3. PMID 31797095
- [Result] Beara-Lasic L, Cogal A, Mara K, Enders F, Mehta RA, Haskic Z, Furth SL, Trachtman H, Scheinman SJ, Milliner DS, Goldfarb DS, Harris PC, Lieske JC; investigators of the Rare Kidney Stone Consortium. Prevalence of low molecular weight proteinuria and Dent disease 1 CLCN5 mutations in proteinuric cohorts. Pediatr Nephrol. 2020 Apr;35(4):633-640. doi: 10.1007/s00467-019-04210-0. Epub 2019 Mar 10. PMID 30852663
- [Result] Brady TM, Roem J, Cox C, Schneider MF, Wilson AC, Furth SL, Warady BA, Mitsnefes M. Adiposity, Sex, and Cardiovascular Disease Risk in Children With CKD: A Longitudinal Study of Youth Enrolled in the Chronic Kidney Disease in Children (CKiD) Study. Am J Kidney Dis. 2020 Aug;76(2):166-173. doi: 10.1053/j.ajkd.2020.01.011. Epub 2020 May 7. PMID 32389356
- [Result] Brown DD, Roem J, Ng DK, Reidy KJ, Kumar J, Abramowitz MK, Mak RH, Furth SL, Schwartz GJ, Warady BA, Kaskel FJ, Melamed ML. Low Serum Bicarbonate and CKD Progression in Children. Clin J Am Soc Nephrol. 2020 Jun 8;15(6):755-765. doi: 10.2215/CJN.07060619. Epub 2020 May 28. PMID 32467307
- [Result] Carlson J, Gerson AC, Matheson MB, Manne S, Warady BA, Hooper SR, Lande M, Harshman LA, Johnson RJ, Shinnar S, Kogon AJ, Furth S. A longitudinal analysis of the effect of anemia on health-related quality of life in children with mild-to-moderate chronic kidney disease. Pediatr Nephrol. 2020 Sep;35(9):1659-1667. doi: 10.1007/s00467-020-04569-5. Epub 2020 Apr 24. PMID 32333284
- [Result] Flynn JT, Carroll MK, Ng DK, Furth SL, Warady BA. Achieved clinic blood pressure level and chronic kidney disease progression in children: a report from the Chronic Kidney Disease in Children cohort. Pediatr Nephrol. 2021 Jun;36(6):1551-1559. doi: 10.1007/s00467-020-04833-8. Epub 2020 Nov 16. PMID 33200315
- [Result] Greenberg JH, Abraham AG, Xu Y, Schelling JR, Feldman HI, Sabbisetti VS, Gonzalez MC, Coca S, Schrauben SJ, Waikar SS, Ramachandran VS, Shlipak MG, Warady B, Kimmel PL, Bonventre JV, Denburg M, Parikh CR, Furth S; CKD Biomarkers Consortium. Plasma Biomarkers of Tubular Injury and Inflammation Are Associated with CKD Progression in Children. J Am Soc Nephrol. 2020 May;31(5):1067-1077. doi: 10.1681/ASN.2019070723. Epub 2020 Mar 31. PMID 32234829
- [Result] Harshman LA, Kogon AJ, Matheson MB, Johnson RJ, Shinnar S, Gerson AC, Warady BA, Furth SL, Hooper SR, Lande MB. Bicarbonate, blood pressure, and executive function in pediatric CKD-is there a link? Pediatr Nephrol. 2020 Jul;35(7):1323-1330. doi: 10.1007/s00467-020-04507-5. Epub 2020 Apr 15. PMID 32297000
- [Result] Hogan J, Schneider MF, Pai R, Denburg MR, Kogon A, Brooks ER, Kaskel FJ, Reidy KJ, Saland JM, Warady BA, Furth SL, Patzer RE, Greenbaum LA. Grip strength in children with chronic kidney disease. Pediatr Nephrol. 2020 May;35(5):891-899. doi: 10.1007/s00467-019-04461-x. Epub 2020 Jan 13. PMID 31932960
- [Result] Jacobson MH, Liu M, Wu Y, Furth S, Warady B, Trachtman H, Trasande L. Oxidant stress and renal function among children with chronic kidney disease: a repeated measures study. Sci Rep. 2020 Feb 21;10(1):3129. doi: 10.1038/s41598-020-59962-9. PMID 32081951
- [Result] Jacobson MH, Wu Y, Liu M, Attina TM, Naidu M, Karthikraj R, Kannan K, Warady BA, Furth S, Vento S, Trachtman H, Trasande L. Serially assessed bisphenol A and phthalate exposure and association with kidney function in children with chronic kidney disease in the US and Canada: A longitudinal cohort study. PLoS Med. 2020 Oct 14;17(10):e1003384. doi: 10.1371/journal.pmed.1003384. eCollection 2020 Oct. PMID 33052911
- [Result] Johnson RJ, Gerson AC, Harshman LA, Matheson MB, Shinnar S, Lande MB, Kogon A, Gipson DS, Warady BA, Furth SL, Hooper SR. A longitudinal examination of parent-reported emotional-behavioral functioning of children with mild to moderate chronic kidney disease. Pediatr Nephrol. 2020 Jul;35(7):1287-1295. doi: 10.1007/s00467-020-04511-9. Epub 2020 Mar 10. PMID 32157444
- [Result] Kim HS, Ng DK, Matheson MB, Atkinson MA, Warady BA, Furth SL, Ruebner RL. Delayed menarche in girls with chronic kidney disease and the association with short stature. Pediatr Nephrol. 2020 Aug;35(8):1471-1475. doi: 10.1007/s00467-020-04559-7. Epub 2020 Apr 27. PMID 32337637
- [Result] Kupferman JC, Matheson MB, Lande MB, Flynn JT, Furth S, Warady BA, Hooper SR. Increased history of ischemic stroke and decreased neurocognitive performance in children with chronic kidney disease. Pediatr Nephrol. 2020 Jul;35(7):1315-1321. doi: 10.1007/s00467-020-04503-9. Epub 2020 Feb 24. PMID 32095895
- [Result] Laster M, Denburg M, Okuda Y, Kumar J, Furth S, Warady B, Kalantar-Zadeh K, Norris K, Salusky IB. Race and Ethnicity Predict Bone Markers and Fracture in Pediatric Patients With Chronic Kidney Disease. J Bone Miner Res. 2021 Feb;36(2):298-304. doi: 10.1002/jbmr.4182. Epub 2020 Oct 23. PMID 32960469
- [Result] Lee J, McCulloch CE, Flynn JT, Samuels J, Warady BA, Furth SL, Seth D, Grimes BA, Mitsnefes MM, Ku E. Prognostic Value of Ambulatory Blood Pressure Load in Pediatric CKD. Clin J Am Soc Nephrol. 2020 Apr 7;15(4):493-500. doi: 10.2215/CJN.10130819. Epub 2020 Mar 11. PMID 32160993
- [Result] Madueme PC, Ng DK, Guju L, Longshore L, Moore V, Jefferies L, Warady BA, Furth S, Mitsnefes M. Aortic dilatation in children with mild to moderate chronic kidney disease. Pediatr Nephrol. 2020 Jun;35(6):1023-1031. doi: 10.1007/s00467-019-04469-3. Epub 2020 Jan 15. PMID 31940069
- [Result] McLeod DJ, Sebastiao YV, Ching CB, Greenberg JH, Furth SL, Becknell B. Longitudinal kidney injury biomarker trajectories in children with obstructive uropathy. Pediatr Nephrol. 2020 Oct;35(10):1907-1914. doi: 10.1007/s00467-020-04602-7. Epub 2020 May 22. PMID 32444926
- [Result] Ng DK, Antiporta DA, Matheson MB, Munoz A. Nonparametric Assessment of Differences Between Competing Risk Hazard Ratios: Application to Racial Differences in Pediatric Chronic Kidney Disease Progression. Clin Epidemiol. 2020 Jan 20;12:83-93. doi: 10.2147/CLEP.S225763. eCollection 2020. PMID 32021474
- [Result] Ng DK, Xu Y, Hogan J, Saland JM, Greenbaum LA, Furth SL, Warady BA, Wong CS. Timing of patient-reported renal replacement therapy planning discussions by disease severity among children and young adults with chronic kidney disease. Pediatr Nephrol. 2020 Oct;35(10):1925-1933. doi: 10.1007/s00467-020-04542-2. Epub 2020 May 3. PMID 32363486
- [Result] Pierce CB, Munoz A, Ng DK, Warady BA, Furth SL, Schwartz GJ. Age- and sex-dependent clinical equations to estimate glomerular filtration rates in children and young adults with chronic kidney disease. Kidney Int. 2021 Apr;99(4):948-956. doi: 10.1016/j.kint.2020.10.047. Epub 2020 Dec 8. PMID 33301749
- [Result] Reynolds BC, Roem JL, Ng DKS, Matsuda-Abedini M, Flynn JT, Furth SL, Warady BA, Parekh RS. Association of Time-Varying Blood Pressure With Chronic Kidney Disease Progression in Children. JAMA Netw Open. 2020 Feb 5;3(2):e1921213. doi: 10.1001/jamanetworkopen.2019.21213. PMID 32058554
- [Result] Schneider MF, Munoz A, Ku E, Warady BA, Furth SL, Schwartz GJ. Estimation of Albumin-Creatinine Ratio From Protein-Creatinine Ratio in Urine of Children and Adolescents With CKD. Am J Kidney Dis. 2021 May;77(5):824-827. doi: 10.1053/j.ajkd.2020.07.015. Epub 2020 Sep 6. No abstract available. PMID 32898620
- [Result] Weidemann DK, Abraham AG, Roem JL, Furth SL, Warady BA. Plasma Soluble Urokinase Plasminogen Activator Receptor (suPAR) and CKD Progression in Children. Am J Kidney Dis. 2020 Aug;76(2):194-202. doi: 10.1053/j.ajkd.2019.11.004. Epub 2020 Jan 24. PMID 31987488
- [Result] Yokoyama JS, Matsuda-Abedini M, Denburg MR, Kumar J, Warady BA, Furth SL, Hooper SR, Portale AA, Perwad F. Association Between Chronic Kidney Disease-Mineral Bone Disease (CKD-MBD) and Cognition in Children: Chronic Kidney Disease in Children (CKiD) Study. Kidney Med. 2020 May 26;2(4):398-406. doi: 10.1016/j.xkme.2020.03.005. eCollection 2020 Jul-Aug. PMID 32775979
- [Result] Abraham AG, Xu Y, Roem JL, Greenberg JH, Weidemann DK, Sabbisetti VS, Bonventre JV, Denburg M, Warady BA, Furth SL. Variability in CKD Biomarker Studies: Soluble Urokinase Plasminogen Activator Receptor (suPAR) and Kidney Disease Progression in the Chronic Kidney Disease in Children (CKiD) Study. Kidney Med. 2021 Jun 17;3(5):712-721.e1. doi: 10.1016/j.xkme.2021.04.007. eCollection 2021 Sep-Oct. PMID 34693253
- [Result] Atkinson MA, Ng DK, Warady BA, Furth SL, Flynn JT. The CKiD study: overview and summary of findings related to kidney disease progression. Pediatr Nephrol. 2021 Mar;36(3):527-538. doi: 10.1007/s00467-019-04458-6. Epub 2020 Feb 3. PMID 32016626
- [Result] Denburg MR, Xu Y, Abraham AG, Coresh J, Chen J, Grams ME, Feldman HI, Kimmel PL, Rebholz CM, Rhee EP, Vasan RS, Warady BA, Furth SL; CKD Biomarkers Consortium. Metabolite Biomarkers of CKD Progression in Children. Clin J Am Soc Nephrol. 2021 Aug;16(8):1178-1189. doi: 10.2215/CJN.00220121. PMID 34362785
- [Result] Diaz-Gonzalez de Ferris ME, Pierce CB, Gipson DS, Furth SL, Warady BA, Hooper SR; Authoring group for the CKiD Study. Health-related quality of life in children with chronic kidney disease is affected by the number of medications. Pediatr Nephrol. 2021 May;36(5):1307-1310. doi: 10.1007/s00467-021-04919-x. Epub 2021 Feb 5. PMID 33547529
- [Result] Dionne JM, Jiang S, Ng DK, Flynn JT, Mitsnefes MM, Furth SL, Warady BA, Samuels JA; CKiD study group. Mean Arterial Pressure and Chronic Kidney Disease Progression in the CKiD Cohort. Hypertension. 2021 Jul;78(1):65-73. doi: 10.1161/HYPERTENSIONAHA.120.16692. Epub 2021 Jun 1. PMID 34058856
- [Result] Greenberg JH, Abraham AG, Xu Y, Schelling JR, Feldman HI, Sabbisetti VS, Ix JH, Jogalekar MP, Coca S, Waikar SS, Shlipak MG, Warady BA, Vasan RS, Kimmel PL, Bonventre JV, Denburg M, Parikh CR, Furth S; CKD Biomarkers Consortium; CKD Biomarker consortium. Urine Biomarkers of Kidney Tubule Health, Injury, and Inflammation are Associated with Progression of CKD in Children. J Am Soc Nephrol. 2021 Oct;32(10):2664-2677. doi: 10.1681/ASN.2021010094. Epub 2021 Sep 20. PMID 34544821
- [Result] Harrell W, Gipson DS, Belger A, Matsuda-Abedini M, Bjornson B, Hooper SR. Functional Magnetic Resonance Imaging Findings in Children and Adolescents With Chronic Kidney Disease: Preliminary Findings. Semin Nephrol. 2021 Sep;41(5):462-475. doi: 10.1016/j.semnephrol.2021.09.009. PMID 34916008
- [Result] Hooper SR, Johnson RJ, Gerson AC, Lande MB, Shinnar S, Harshman LA, Kogon AJ, Matheson M, Bartosh S, Carlson J, Warady BA, Furth SL. Overview of the findings and advances in the neurocognitive and psychosocial functioning of mild to moderate pediatric CKD: perspectives from the Chronic Kidney Disease in Children (CKiD) cohort study. Pediatr Nephrol. 2022 Apr;37(4):765-775. doi: 10.1007/s00467-021-05158-w. Epub 2021 Jun 10. PMID 34110493
- [Result] Hooper SR, Johnson RJ, Lande M, Matheson M, Shinnar S, Kogon AJ, Harshman L, Spinale J, Gerson AC, Warady BA, Furth SL. The Similarities and Differences Between Glomerular vs. Non-glomerular Diagnoses on Intelligence and Executive Functions in Pediatric Chronic Kidney Disease: A Brief Report. Front Neurol. 2021 Dec 20;12:787602. doi: 10.3389/fneur.2021.787602. eCollection 2021. PMID 34987470
- [Result] Jacobson MH, Wu Y, Liu M, Kannan K, Li AJ, Robinson M, Warady BA, Furth S, Trachtman H, Trasande L. Organophosphate pesticides and progression of chronic kidney disease among children: A prospective cohort study. Environ Int. 2021 Oct;155:106597. doi: 10.1016/j.envint.2021.106597. Epub 2021 May 2. PMID 33951537
- [Result] Kim HS, Ng DK, Matheson MB, Atkinson MA, Akhtar Y, Warady BA, Furth SL, Ruebner RL. Association of Puberty With Changes in GFR in Children With CKD. Am J Kidney Dis. 2022 Jan;79(1):131-134. doi: 10.1053/j.ajkd.2021.05.011. Epub 2021 Jun 24. No abstract available. PMID 34171395
- [Result] Levy RV, Reidy KJ, Le TH, David V, Winkler C, Xu Y, Warady B, Furth S, Kaskel F, Melamed ML. Association of GSTM1 Deletion With Progression of CKD in Children: Findings From the Chronic Kidney Disease in Children (CKiD) Study. Am J Kidney Dis. 2022 Jul;80(1):79-86. doi: 10.1053/j.ajkd.2021.10.007. Epub 2021 Dec 4. PMID 34871703
- [Result] Mitsnefes MM, Xu Y, Ng DK, Hill G, Kimball T, Furth SL, Warady BA. Diastolic Function and Ambulatory Hypertension in Children With Chronic Kidney Disease. Hypertension. 2021 Nov;78(5):1347-1354. doi: 10.1161/HYPERTENSIONAHA.121.17449. Epub 2021 Oct 4. PMID 34601967
- [Result] Molino AR, Jerry-Fluker J, Atkinson MA, Furth SL, Warady BA, Ng DK. Alcohol, cigarette, e-cigarette and marijuana use among adolescents and young adults with chronic kidney disease in North America. Ann Epidemiol. 2021 Jul;59:56-63. doi: 10.1016/j.annepidem.2021.04.001. Epub 2021 Apr 22. PMID 33894386
- [Result] Molino AR, Jerry-Fluker J, Atkinson MA, Furth SL, Warady BA, Ng DK. The association of alcohol, cigarette, e-cigarette, and marijuana use with disease severity in adolescents and young adults with pediatric chronic kidney disease. Pediatr Nephrol. 2021 Aug;36(8):2493-2497. doi: 10.1007/s00467-021-05044-5. Epub 2021 Apr 29. PMID 33914145
- [Result] Ng DK, Carroll MK, Kaskel FJ, Furth SL, Warady BA, Greenbaum LA. Patterns of recombinant growth hormone therapy use and growth responses among children with chronic kidney disease. Pediatr Nephrol. 2021 Dec;36(12):3905-3913. doi: 10.1007/s00467-021-05122-8. Epub 2021 Jun 11. PMID 34115207
- [Result] Ng DK, Furth SL, Warady BA, Crews DC, Seegmiller JC, Schwartz GJ; CKiD Study Investigators. Self-reported Race, Serum Creatinine, Cystatin C, and GFR in Children and Young Adults With Pediatric Kidney Diseases: A Report From the Chronic Kidney Disease in Children (CKiD) Study. Am J Kidney Dis. 2022 Aug;80(2):174-185.e1. doi: 10.1053/j.ajkd.2021.10.013. Epub 2021 Dec 30. PMID 34974031
- [Result] Ng DK, Pierce CB. Kidney Disease Progression in Children and Young Adults With Pediatric CKD: Epidemiologic Perspectives and Clinical Applications. Semin Nephrol. 2021 Sep;41(5):405-415. doi: 10.1016/j.semnephrol.2021.09.002. PMID 34916001
- [Result] Richardson KL, Weaver DJ Jr, Ng DK, Carroll MK, Furth SL, Warady BA, Flynn JT. L-type calcium channel blocker use and proteinuria among children with chronic kidney diseases. Pediatr Nephrol. 2021 Aug;36(8):2411-2419. doi: 10.1007/s00467-021-04967-3. Epub 2021 Feb 15. PMID 33590332
- [Result] Rodig NM, Roem J, Schneider MF, Seo-Mayer PW, Reidy KJ, Kaskel FJ, Kogon AJ, Furth SL, Warady BA. Longitudinal outcomes of body mass index in overweight and obese children with chronic kidney disease. Pediatr Nephrol. 2021 Jul;36(7):1851-1860. doi: 10.1007/s00467-020-04907-7. Epub 2021 Jan 21. PMID 33479822
- [Result] Sandokji I, Greenberg JH. Plasma and Urine Biomarkers of CKD: A Review of Findings in the CKiD Study. Semin Nephrol. 2021 Sep;41(5):416-426. doi: 10.1016/j.semnephrol.2021.09.003. PMID 34916002
- [Result] Sgambat K, Roem J, Brady TM, Flynn JT, Mitsnefes M, Samuels JA, Warady BA, Furth SL, Moudgil A. Social Determinants of Cardiovascular Health in African American Children With CKD: An Analysis of the Chronic Kidney Disease in Children (CKiD) Study. Am J Kidney Dis. 2021 Jul;78(1):66-74. doi: 10.1053/j.ajkd.2020.11.013. Epub 2021 Jan 5. PMID 33418013
- [Result] Shah LN, Matheson MB, Furth SL, Schwartz GJ, Warady BA, Wong CJ. Low variability of plant protein intake in the CKiD cohort does not demonstrate changes in estimated GFR nor electrolyte balance. Pediatr Nephrol. 2022 Jul;37(7):1647-1655. doi: 10.1007/s00467-021-05334-y. Epub 2021 Nov 18. PMID 34796391
- [Result] Verbitsky M, Krithivasan P, Batourina E, Khan A, Graham SE, Marasa M, Kim H, Lim TY, Weng PL, Sanchez-Rodriguez E, Mitrotti A, Ahram DF, Zanoni F, Fasel DA, Westland R, Sampson MG, Zhang JY, Bodria M, Kil BH, Shril S, Gesualdo L, Torri F, Scolari F, Izzi C, van Wijk JAE, Saraga M, Santoro D, Conti G, Barton DE, Dobson MG, Puri P, Furth SL, Warady BA, Pisani I, Fiaccadori E, Allegri L, Degl'Innocenti ML, Piaggio G, Alam S, Gigante M, Zaza G, Esposito P, Lin F, Simoes-E-Silva AC, Brodkiewicz A, Drozdz D, Zachwieja K, Miklaszewska M, Szczepanska M, Adamczyk P, Tkaczyk M, Tomczyk D, Sikora P, Mizerska-Wasiak M, Krzemien G, Szmigielska A, Zaniew M, Lozanovski VJ, Gucev Z, Ionita-Laza I, Stanaway IB, Crosslin DR, Wong CS, Hildebrandt F, Barasch J, Kenny EE, Loos RJF, Levy B, Ghiggeri GM, Hakonarson H, Latos-Bielenska A, Materna-Kiryluk A, Darlow JM, Tasic V, Willer C, Kiryluk K, Sanna-Cherchi S, Mendelsohn CL, Gharavi AG. Copy Number Variant Analysis and Genome-wide Association Study Identify Loci with Large Effect for Vesicoureteral Reflux. J Am Soc Nephrol. 2021 Apr;32(4):805-820. doi: 10.1681/ASN.2020050681. Epub 2021 Feb 17. PMID 33597122
- [Result] Viteri B, Elsingergy M, Roem J, Ng D, Warady B, Furth S, Tasian G. Ultrasound-Based Renal Parenchymal Area and Kidney Function Decline in Infants With Congenital Anomalies of the Kidney and Urinary Tract. Semin Nephrol. 2021 Sep;41(5):427-433. doi: 10.1016/j.semnephrol.2021.09.004. PMID 34916003
- [Result] Xu Y, Ng DK, Furth SL, Warady BA, Mitsnefes MM. Factors associated with the absence of pharmacological treatment for common modifiable complications in children with chronic kidney disease. Pediatr Nephrol. 2021 Oct;36(10):3181-3189. doi: 10.1007/s00467-021-05087-8. Epub 2021 May 6. PMID 33959814
- [Result] Johnson RJ, Harshman LA. Neurocognition in Pediatric Chronic Kidney Disease: A Review of Data From the Chronic Kidney Disease in Children (CKiD) Study. Semin Nephrol. 2021 Sep;41(5):446-454. doi: 10.1016/j.semnephrol.2021.09.007. PMID 34916006
- [Result] Akchurin O, Molino AR, Schneider MF, Atkinson MA, Warady BA, Furth SL. Longitudinal Relationship Between Anemia and Statural Growth Impairment in Children and Adolescents With Nonglomerular CKD: Findings From the Chronic Kidney Disease in Children (CKiD) Study. Am J Kidney Dis. 2023 Apr;81(4):457-465.e1. doi: 10.1053/j.ajkd.2022.09.019. Epub 2022 Dec 5. PMID 36481700
- [Result] Bakhoum CY, Katz R, Samuels JA, Al-Rousan T, Furth SL, Ix JH, Garimella PS. Nocturnal Dipping and Left Ventricular Mass Index in the Chronic Kidney Disease in Children Cohort. Clin J Am Soc Nephrol. 2022 Jan;17(1):75-82. doi: 10.2215/CJN.09810721. Epub 2021 Nov 12. PMID 34772729
- [Result] Bakhoum CY, Matheson MB, Greenberg JH, Furth SL, Ix JH, Garimella PS. Urine Uromodulin Is Not Associated With Blood Pressure in the Chronic Kidney Disease in Children Cohort. Hypertension. 2022 Oct;79(10):2298-2304. doi: 10.1161/HYPERTENSIONAHA.122.19566. Epub 2022 Aug 3. PMID 35920156
- [Result] Bakhoum CY, Phadke M, Deng Y, Samuels JA, Garimella PS, Furth SL, Wilson FP, Ix JH. Nocturnal Dipping and Kidney Function Decline: Findings From the CKD in Children Study. Kidney Int Rep. 2022 Aug 17;7(11):2446-2453. doi: 10.1016/j.ekir.2022.08.002. eCollection 2022 Nov. PMID 36531891
- [Result] Boynton SA, Matheson MB, Ng DK, Hidalgo G, Warady BA, Furth SL, Atkinson MA. The Relationship Between Neighborhood Disadvantage and Kidney Disease Progression in the Chronic Kidney Disease in Children (CKiD) Cohort. Am J Kidney Dis. 2022 Aug;80(2):207-214. doi: 10.1053/j.ajkd.2021.12.008. Epub 2022 Jan 25. PMID 35085688
- [Result] Guzman-Limon ML, Jiang S, Ng D, Flynn JT, Warady B, Furth SL, Samuels JA; Chronic Kidney Disease in Children study*. Nocturnal Hypertension in Children With Chronic Kidney Disease Is Common and Associated With Progression to Kidney Replacement Therapy. Hypertension. 2022 Oct;79(10):2288-2297. doi: 10.1161/HYPERTENSIONAHA.121.18101. Epub 2022 Aug 18. PMID 35979846
- [Result] Jacobson MH, Wu Y, Liu M, Kannan K, Lee S, Ma J, Warady BA, Furth S, Trachtman H, Trasande L. Urinary Polycyclic Aromatic Hydrocarbons in a Longitudinal Cohort of Children with CKD: A Case of Reverse Causation? Kidney360. 2022 Mar 29;3(6):1011-1020. doi: 10.34067/KID.0000892022. eCollection 2022 Jun 30. PMID 35845343
- [Result] Kogon AJ, Roem J, Schneider MF, Mitsnefes MM, Zemel BS, Warady BA, Furth SL, Rodig NM. Associations of body mass index (BMI) and BMI change with progression of chronic kidney disease in children. Pediatr Nephrol. 2023 Apr;38(4):1257-1266. doi: 10.1007/s00467-022-05655-6. Epub 2022 Aug 26. PMID 36018433
- [Result] Lee AM, Hu J, Xu Y, Abraham AG, Xiao R, Coresh J, Rebholz C, Chen J, Rhee EP, Feldman HI, Ramachandran VS, Kimmel PL, Warady BA, Furth SL, Denburg MR; CKD Biomarkers Consortium. Using Machine Learning to Identify Metabolomic Signatures of Pediatric Chronic Kidney Disease Etiology. J Am Soc Nephrol. 2022 Feb;33(2):375-386. doi: 10.1681/ASN.2021040538. Epub 2022 Jan 11. PMID 35017168
- [Result] Molino AR, Minnick MLG, Jerry-Fluker J, Karita Muiru J, Boynton SA, Furth SL, Warady BA, Ng DK; Chronic Kidney Disease in Children Study. Health and Dental Insurance and Health Care Utilization Among Children, Adolescents, and Young Adults With CKD: Findings From the CKiD Cohort Study. Kidney Med. 2022 Mar 25;4(5):100455. doi: 10.1016/j.xkme.2022.100455. eCollection 2022 May. PMID 35518833
- [Result] Ng DK, Carroll MK, Furth SL, Warady BA, Flynn JT; CKiD Study Investigators. Blood Pressure Classification Status in Children With CKD Following Adoption of the 2017 American Academy of Pediatrics Guideline. Am J Kidney Dis. 2023 May;81(5):545-553. doi: 10.1053/j.ajkd.2022.10.009. Epub 2022 Dec 12. PMID 36521780
- [Result] Schwartz GJ, Roem JL, Hooper SR, Furth SL, Weaver DJ Jr, Warady BA, Schneider MF. Longitudinal changes in uric acid concentration and their relationship with chronic kidney disease progression in children and adolescents. Pediatr Nephrol. 2023 Feb;38(2):489-497. doi: 10.1007/s00467-022-05620-3. Epub 2022 Jun 1. PMID 35650320
- [Result] Bae S, Samuels JA, Flynn JT, Mitsnefes MM, Furth SL, Warady BA, Ng DK; CKiD Study. Machine Learning-Based Prediction of Masked Hypertension Among Children With Chronic Kidney Disease. Hypertension. 2022 Sep;79(9):2105-2113. doi: 10.1161/HYPERTENSIONAHA.121.18794. Epub 2022 Jul 7. PMID 35862083
- [Result] Brown DD, Carroll M, Ng DK, Levy RV, Greenbaum LA, Kaskel FJ, Furth SL, Warady BA, Melamed ML, Dauber A. Longitudinal Associations between Low Serum Bicarbonate and Linear Growth in Children with CKD. Kidney360. 2022 Feb 9;3(4):666-676. doi: 10.34067/KID.0005402021. eCollection 2022 Apr 28. PMID 35721607
- [Result] Douglas CE, Roem J, Flynn JT, Furth SL, Warady BA, Halbach SM; Chronic Kidney Disease in Children study investigators*. Effect of Age on Hypertension Recognition in Children With Chronic Kidney Disease: A Report From the Chronic Kidney Disease in Children Study. Hypertension. 2023 May;80(5):1048-1056. doi: 10.1161/HYPERTENSIONAHA.122.20354. Epub 2023 Mar 2. PMID 36861464
- [Result] Bae S, Schwartz GJ, Mendley SR, Warady BA, Furth SL, Munoz A; CKiD Study Investigators. Trajectories of eGFR after kidney transplantation according to trajectories of eGFR prior to kidney replacement therapies in children with chronic kidney disease. Pediatr Nephrol. 2023 Dec;38(12):4157-4164. doi: 10.1007/s00467-023-06056-z. Epub 2023 Jun 23. PMID 37353626
- [Result] Carlson J, Gerson AC, Matheson MB, Manne S, Lande M, Harshman L, Johnson RJ, Shinnar S, Kogon AJ, Warady B, Furth S, Hooper S. Longitudinal changes of health-related quality of life in childhood chronic kidney disease. Pediatr Nephrol. 2023 Dec;38(12):4127-4136. doi: 10.1007/s00467-023-06069-8. Epub 2023 Jul 10. PMID 37428223
- [Result] Faulkner SC, Matheson MB, Greenberg JH, Garimella PS, Furth SL, Ix JH, Bakhoum CY. Association of clinical characteristics with urine uromodulin in children with chronic kidney disease. Pediatr Nephrol. 2023 Nov;38(11):3859-3862. doi: 10.1007/s00467-023-05947-5. Epub 2023 Mar 29. PMID 36988691
- [Result] Harshman LA, Ward RC, Matheson MB, Dawson A, Kogon AJ, Lande MB, Molitor SJ, Johnson RJ, Wilson C, Warady BA, Furth SL, Hooper SR. The Impact of Pediatric CKD on Educational and Employment Outcomes. Kidney360. 2023 Oct 1;4(10):1389-1396. doi: 10.34067/KID.0000000000000206. Epub 2023 Jul 7. PMID 37418621
- [Result] Kula AJ, Flynn JT, Prince DK, Furth SL, Warady B, Isakova T, Christenson R, Bansal N. Descriptions and Determinants of N-Terminal Pro-B-Type Natriuretic Peptide in Pediatric CKD: The Chronic Kidney Disease in Children (CKiD) Study. Am J Kidney Dis. 2023 Dec;82(6):776-778. doi: 10.1053/j.ajkd.2023.03.020. Epub 2023 Jun 29. No abstract available. PMID 37393051
- See also: CKiD Website — https://statepi.jhsph.edu/ckid/